CLINICAL TRIAL: NCT04851106
Title: Evaluation of Endoscopic Ultrasound Shear Wave Elastography (EUS-SWE) for the Diagnosis of Pancreatic Adenocarcinoma.
Acronym: EDEN
Status: Recruiting | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A02679-30
Record Dates: First submitted 2021-04-15; First posted 2021-04-20 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Endosonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with a solid pancreatic lesion of an undetermined nature: Patient with a solid pancreatic lesion of an undetermined nature
  Interventions: Diagnostic Test: Endoscopic ultrasound

INTERVENTIONS:
Diagnostic Test: Endoscopic ultrasound — Diagnosis of pancreatic adenocarcinoma with endoscopic ultrasound.

SUMMARY:
To assess the diagnostic accuracy of Shear Wave elastography (SWE) for the diagnosis of pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
Pancreatic adenocarcinoma (PA) is the most common tumor of the pancreas, representing more than 90% of all solid pancreatic neoplasia and 55% -73% of solid pancreatic masses.

Given its poor prognosis and the major therapeutic consequences, the discrimination between PA and other pancreatic solid lesions is mandatory. Endoscopic ultrasound (EUS) is admitted as the most sensitive imaging procedure for the detection and characterization of pancreatic tumors. Based on only endosonographic features, it remains difficult to differentiate PA from other solid masses, the specificity (Spe) and accuracy of EUS for the diagnosis of pancreatic tumor malignancy range from 53-69% and 72-83%, respectively. Over the last 15 years, endoscopic ultrasound fine needle aspiration (EUS-FNA) or more recently fine needle biopsy (EUS-FNB) has demonstrated its efficiency for tissue sampling and pathologic diagnosis of PA. Complementary techniques have been developed to increase the diagnostic performance of EUS. EUS-Elastography (EUS-E) is another EUS image enhancement technique, which rational based on the difference in elasticity between the tissues. There are two types of elastographies: strain elastography (SE) and shear wave elastography (SWE).

Several studies have demonstrated the utility of ultrasound SWE (US-SWE) for the differential diagnosis of lesions of the breast, thyroid, prostate and for detection of pancreatic fibrosis and chronic pancreatitis. However, to date, there is no data about the performance of EUS-SWE for the differential diagnosis of pancreatic solid lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Patient with a solid pancreatic mass of indeterminate origin

Exclusion Criteria:

* Patient with ASA score 4 or 5
* Patient with contraindication to SonoVue injection
* Protected patient : major under guardianship, tutorship or other legal protection, deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with a solid pancreatic mass of indeterminate origin
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2021-09-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The negative predictive value (NPV) determined from shear wave elastography | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rodica GINCUL, Principal Investigator — Hôpital Jean Mermoz
Locations (1):
- Hôpital Jean Mermoz, Lyon, France

IPD SHARING:
Plan to Share IPD: No